CLINICAL TRIAL: NCT05858385
Title: Risk Prediction of Severe Radiation-induced Oral Mucositis in Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Predictive Study on Acute Radiation Induced Oral Mucositis in Nasopharyngeal Carcinoma Patients
Status: Recruiting | Type: Observational
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: oral mucositis
Record Dates: First submitted 2023-04-20; First posted 2023-05-15 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Nasopharyngeal Carcinoma by AJCC V8 Stage; Radiation Induced Mucositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Development and Validation of severe RIOM prediction model: This group aims to develop an artificial intelligence model using a retrospective cohort to predict severe RIOM in patients diagnosed with LA-NPC and evaluate risk factors for severe RIOM and further validate the effectiveness of this risk factor in reducing the risk of severe RIOM on risk factors for severe RIOM identified by the predictive model.The oral evaluation of all patients was conducted by the same senior dentist, who evaluated the oral mucosal radiation toxicity weekly at baseline (before RT) and after RT, and performed RIOM scores.RIOM is classified using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v5.0) .
  Interventions: Other: Intervention based on key factors identified by the severe RIOM prediction model

INTERVENTIONS:
Other: Intervention based on key factors identified by the severe RIOM prediction model — Intervention based on key factors identified by the severe RIOM prediction model

SUMMARY:
Exploring effective risk prediction models for severe Radiation-Induced Oral Mucositis (RIOM/RTOM), providing a research basis for mitigating oral radiation toxicity, and effectively improving the sensitivity of dentists in predicting the risk of severe RIOM in locally advanced nasopharyngeal carcinoma patients.Based on precise radiotherapy, it is proposed to extract OAR using the contour of local oral areas. Explore more accurate RIOM dose-response relationships.Exploring a new type of fusion classifier, by complementing the information between each base classifier, helps to maximize the utilization of the information contained in different factors to build a more objective, reliable, and efficient multi criteria decision-making based risk prediction model for severe RIOM. It use predictive models to identify key risk factors for severe RIOM and further validate the effectiveness of this risk factor in reducing the risk of severe RIOM on risk factors for severe RIOM identified by the predictive mode.

DETAILED DESCRIPTION:
This study investigates the prediction and management of Radiation-Induced Oral Mucositis (RIOM/RTOM) in patients with locally advanced nasopharyngeal carcinoma undergoing radiotherapy. RIOM is a significant concern due to its impact on the quality of life for patients and its potential to disrupt radiotherapy courses, affecting local tumor control rates. We systematically analyzed multifaceted data, including dosimetric parameters, clinical factors, and oral variables, to develop a predictive model for severe RIOM. The effectiveness of key risk factors in mitigating the risk of severe RIOM was further validated to predict and potentially prevent severe RIOM.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed as nasopharyngeal carcinoma through pathological tissue biopsy, AJCC 8th edition bed staging is I-Iva stage, with no distant metastasis
* First time receiving radical radiation therapy and receiving RTOM observation and treatment throughout the entire process in the Department of Stomatology
* Complete information on anti-tumor treatment materials
* No oral mucosal diseases that have not been effectively controlled in the past or still require long-term medication treatment
* Other diseases that do not affect the treatment of nasopharyngeal carcinoma

Exclusion Criteria:

* Failure to complete radiotherapy, or material release time delayed by more than two weeks compared to plan
* There are other diseases that affect the examination and treatment of oral mucosal inflammation, such as restricted mouth opening, Schegren's syndrome, etc
* Expected survival time less than 6 months
* Cases where patients withdraw from clinical trials at any time and for any reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nasopharyngeal cancer patients diagnosed with tissue biopsy and no distant metastasis, who underwent RTOM observation and treatment throughout the radiotherapy period in the Department of Stomatology
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe RIOM | during radiotherapy
  According to the CTCAE V5.0 ，Grade 3 and Grade 4 is considered severe RTOM

SECONDARY OUTCOMES:
Risk factors of severe RIOM | baseline (before radiotherapy)
  Patient factors, disease factors, and treatment related factors

OTHER OUTCOMES:
Changes from oral dryness in RIOM patients | Baseline, the 10th, 20th and 30th days of radiotherapy
  According to the Clinical oral dryness score(CODS),A total of 10 features were used to obtain the total CODS. A high total score indicates increased oral dryness.
Changes from salivary PH compared to baseline in RIOM patients | Baseline, the 10th, 20th and 30th days of radiotherapy
  Evaluation of salivary PH using pH indicator paper
Changes from the pain in xerostomia combined with RIOM patients | Baseline, the 10th, 20th and 30th days of radiotherapy
  The evaluation of pain is based on the Numerical Rating Scale (NRS), with a numerical score of 0-10. A score of less than 5 is considered mild pain, a score of 5-7 is moderate pain, and a score of 8 or above is severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Yu Zeng, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeng Y, Hu Y, Wang L, Liao Z, Tan J, Kuang Y, Gong P, Qi B, Zhen X. Control of dental calculus Prevents severe Radiation-Induced oral mucositis in patients undergoing radiotherapy for nasopharyngeal carcinoma. Radiother Oncol. 2025 Jun;207:110872. doi: 10.1016/j.radonc.2025.110872. Epub 2025 Mar 27. PMID 40157544